CLINICAL TRIAL: NCT07393607
Title: Acute Effects of Partial Sleep Deprivation on Appetite, Energy Intake and Physical Activity
Brief Title: Effects of Acute Sleep Deprivation on Human Behaviours
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202412HM033-2
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Physical Activity; Energy Intake; Appetite; Food Choice
Keywords: Physical activity; Energy intake; Appetite; Food choice
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep (Experimental): Participants will have an 8-hour sleep opportunity in the lab from 23:00 to 07:00.
  Interventions: Behavioral: Normal sleep
- Partial sleep deprivation (Experimental): Participants will have a 3-hour sleep opportunity in the lab from 03:00 to 07:00.
  Interventions: Behavioral: Partial sleep deprivation

INTERVENTIONS:
Behavioral: Normal sleep — Participants will have an 8-hour sleep opportunity in the lab from 23:00 to 07:00.
  Arms: Normal sleep
Behavioral: Partial sleep deprivation — Participants will have a 3-hour sleep opportunity in the lab from 03:00 to 07:00.
  Arms: Partial sleep deprivation

SUMMARY:
This study will investigate whether acute sleep deprivation affects appetite, eating behavior, and physical activity in both regular exercisers and physically inactive individuals.

DETAILED DESCRIPTION:
Prior to the main trials, participants will complete assessments of V̇O2max and maximal muscle strength within 7 to 14 days before the main trials. They will also record one week of daily physical activity, sleep patterns, and diet (including two weekdays and one weekend day) to ensure they meet the inclusion criteria.

Participants will be healthy males aged 20 to 45, grouped according to their habitual activity levels.

1. Sedentary: fewer than 7,000 steps/day, no regular exercise in the past 6 months.
2. Regular Aerobic Exercise: Running or cycling at least 2-3 times/week for the past 6 months.
3. Regular Resistance Exercise: Engaging in resistance exercise at least 2-3 times/week for the past 6 months, with minimal aerobic training.

Day 1:

Physical activity is restricted to a minimum, with no exercise permitted. Participants are allowed to eat freely before 15:00; however, all food intake will be recorded to enable replication prior to the subsequent main trial. Napping is not permitted. Participants will arrive at the laboratory between 18:30 and 19:00. Subjective appetite sensations and food preferences will be assessed. Participants will have either an 8-hour sleep opportunity in the laboratory from 23:00 to 07:00 (i.e., normal sleep trial) or a 3-hour sleep opportunity from 03:00 to 07:00 (i.e., partial sleep deprivation trial).

Day 2:

Participants will wake at 07:00. After completing personal hygiene, they will rest for 20 minutes to ensure full alertness. At 07:30, a 20-minute resting metabolic rate assessment will be conducted, alongside the collection of heart rate variability and muscle oxygen saturation data. Subsequently, pulse wave velocity measurement, cognitive function tests, subjective questionnaires, and a computerized food preference test will be administered.

After the baseline assessment, a 3-hour oral glucose tolerance test (OGTT) will be administered. Visual analogue scale assessments-including sleep, appetite, and mood-will be conducted every 30 minutes during the OGTT. Food preferences will be measured 180 minutes after the completion of the OGTT. Upon leaving the laboratory, participants will be provided with a pedometer and wearable devices and instructed to record dietary intake (using a food scale and photographic records), sleep, and glucose values on the experimental day and for the following four consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 45 years.
* Body Mass Index (BMI) between 18.5 to 27 kg/m².
* No sleep-related medical conditions and good sleep quality, defined as a Pittsburgh Sleep Quality Index (PSQI) score ≤ 5.
* Usual bedtime between 22:00 and 01:00, wake-up time between 06:00 and 09:00, with an average sleep duration of 7 to 9 hours. Chronotype classified as "definitely not evening type" (score ≥ 42 on the Morningness-Eveningness Questionnaire), with no changes in sleep patterns over the past 3 months.
* Without any metabolic or cardiovascular diseases, and not using medications that could affect metabolic responses.
* No specific dietary habits, such as intermittent fasting or a ketogenic diet.
* Maintaining a stable weight (no self-reported weight change greater than ±3 kg) for at least 3 months.
* Resting blood pressure ≤ 130/80 mmHg.
* No smoking or excessive alcohol consumption.
* Not a shift worker.
* No international travel across time zones in the past 3 months.

Exclusion Criteria:

* Special diets (e.g., intermittent fasting, ketogenic diet)
* Recent injuries or contraindications to intense exercise.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Energy intake | 4 days in a free-living conditions.
  Energy and macronutrients intake will be collected using pictures and via a food scale
Physical activity | 4 days in a free-living conditions.
  Physical activity level and intensity will be collected using wearable devices

SECONDARY OUTCOMES:
Food preference | Baseline and at the end of the 3-hour oral glucose tolerance test (OGTT).
  Computerised subjective food choice
Appetite sensations | At 0 (baseline), 30, 60, 90, 120, 150, and 180 minutes during the 3-hour oral glucose tolerance test (OGTT).
  Subjective appetitive feelings will be measured using a 0-100 mm visual analog scale (VAS), with higher values indicating more intense feelings.
Mood sensations | At 0 (baseline), 30, 60, 90, 120, 150, and 180 minutes during the 3-hour oral glucose tolerance test (OGTT).
  Subjective mood feelings will be measured using a 0-100 mm visual analog scale (VAS), with higher values indicating more intense feelings.
Sleep sensations | At 0 (baseline), 30, 60, 90, 120, 150, and 180 minutes during the 3-hour oral glucose tolerance test (OGTT).
  Subjective sleep feelings will be measured using a 0-100 mm visual analog scale (VAS), with higher values indicating more intense feelings.
Sleep | 4 days in a free-living conditions.
  Sleep duration will be collected via wearable device.
Glucose responses | 4 days in a free-living conditions.
  Clucose responses will be collected using continuous glucose monitoring